CLINICAL TRIAL: NCT05460715
Title: Prospective Multicentre Study to Evaluate the Long-term Performance of Anteverted Femoral Stems in Total Hip Arthroplasty
Brief Title: The Medacta Quadra-P Anteverted Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.001.20
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-03

CONDITIONS: Arthrosis; Traumatic Arthritis; Rheumatoid Polyarthritis; Congenital Hip Dysplasia; Avascular Necrosis of the Femoral Head
Keywords: total hip arthroplasty; Quadra P anteverted; Medacta
MeSH Terms: conditions — Osteoarthritis; Hip Dislocation, Congenital; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: Quadra P anteverted — * Assess clinical performance by Harris Hip score collected during preoperative and postoperative visits at 3 months, 1, 2, 5, 7 and 10 years.
  * Assess radiological performance by standard radiographic examination performed before surgery, after surgery before discharge and during postoperative visits at 3 months, 1, 2, 5, 7 and 10 years.
  * Assessing the patient's perception of the prosthetic joint by means of FJS questionnaire collected during the preoperative visit and postoperative visits at 3 months and at 1, 2, 5, 7 and 10 years after surgery.
  * Assessment of functional recovery by gait analysis study
  * Collect the rate of complications throughout the course of the study

SUMMARY:
This is a Post-Marketing Surveillance of Quadra-P anteverted stem prosthesis.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the 10-year survival of the anteverted Quadra-P stem in patients operated for primary total hip arthroplasty, according to the inclusion criteria.

Secondary objectives:

* To assess clinical performance by Harris Hip score collected during preoperative and postoperative visits at 3 months, 1, 2, 5, 7 and 10 years.
* Assess radiological performance by standard radiographic examination performed preoperatively, postoperatively before discharge and during postoperative visits at 3 months, 1, 2, 5, 7 and 10 years.
* Assessing the patient's perception of the prosthetic joint by means of FJS questionnaire collected during the preoperative visit and postoperative visits at 3 months and at 1, 2, 5, 7 and 10 years after surgery.
* Assessment of functional recovery by gait analysis study
* Collect the rate of complications throughout the course of the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from primary hip arthrosis, post-traumatic arthrosis, dysplasia or avascular necrosis of the femoral head, rheumatoid arthritis
* Adult subjects between 18 and 75 years of age on the date of surgery
* Subjects eligible for primary total hip arthroplasty surgery for whom the anterior Quadra-P femoral component will be implanted according to the indications for use of the implant
* Subjects who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to surgery.

For the anatomical-functional subgroup:

- Adult subjects aged between 18 and 65 years at the date of surgery who have agreed to undergo the gait analysis study.

Exclusion Criteria:

* Subjects with acute or chronic infection
* Subjects with a femoral neck fracture
* Subjects with mental conditions that impair their ability to consent to the study, to complete required questionnaires or to complete follow-up visits
* Subjects with severe deformities, at the discretion of the surgeon
* Subjects with metabolic disorders that may involve bone metabolism for which an uncemented implant would be contraindicated
* Subjects with muscular atrophy or neuromuscular diseases
* Subjects allergic to the materials used during surgery
* Subjects unable or unwilling to provide consent for participation in the study
* Any other condition not mentioned in the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of the study is to monitor the clinical performance and survival of the Quadra-P antevert stem when used according to its indications. Since patients are not subjected to additional risks or procedures compared to standard practice, the total number of patients was defined on the basis of the surgeon's potential and observational studies of the same type already published in the literature.
  For the anatomical-functional subgroup, a sample size was defined to verify 10% speed increases between pre- and postoperative. Considering α = 5% and Power = 90%, 30 patients will be required.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 10-year survival of the anteverted Quadra-P stem | 10 years
  % survival rate

SECONDARY OUTCOMES:
Assess clinical performance | at 3 months, 1, 2, 5, 7 and 10 years.
  Harris Hip score (HHS) (0 minimum-100 maximum)
Assess radiological performance | at pre-op, 3 months, 1, 2, 5, 7 and 10 years.
  Assess radiological performance by standard radiographic examination performed before surgery, after surgery before discharge and during postoperative visits
Assessing the patient's perception of the prosthetic joint | at 3 months and at 1, 2, 5, 7 and 10 years after surgery.
  Forgotten Joint Score (FJS) (0 minimum-100 maximum)
Assessment of functional recovery | at pre-op, 3 months and at 1 year after surgery.
  Assessment of functional recovery by gait analysis study
Collect the rate of complications | at pre-op, immediate post-op, 3 months, 1, 2, 5, 7 and 10 years.
  Collect the rate of complications throughout the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Franco Scalabrino, Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: No